CLINICAL TRIAL: NCT02625467
Title: Treatment of Keratoconus With Pachymetry Assisted Laser Keratoplasty (PALK) Versus Penetrating Keratoplasty (PK)
Brief Title: Treatment of Keratoconus With PALK Versus PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALK vs PK
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Keratoconus
Keywords: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Keratoplasty, Penetrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Penetrating keratoplasty (Experimental): Conventional penetrating keratoplasty technique
  Interventions: Procedure: Penetrating keratoplasty; Drug: Treatment posterior to surgery
- PALK (Experimental): Pachymetry and Excimer laser assisted lamellar keratoplasty
  Interventions: Procedure: Pachymetry and Excimer laser assisted lamellar keratoplasty; Drug: Treatment posterior to surgery

INTERVENTIONS:
Procedure: Penetrating keratoplasty — Conventional Penetrating keratoplasty technique
  Arms: Penetrating keratoplasty
Procedure: Pachymetry and Excimer laser assisted lamellar keratoplasty — Ablation profile focusing on topography and pachymetry with Schwind Amaris excimer laser
  Arms: PALK
Drug: Treatment posterior to surgery — Fluoroquinolone topical antibiotic (Moxifloxacin, Vigamox) and topical steroid (Prednisolone Acetate Ophthalmic Suspension, Pred Forte)

SUMMARY:
The purpose of this study is to evaluate the visual results of patients with keratoconus treated with one of two techniques: penetrating keratoplasty (PK) vs. pachymetry and Excimer laser assisted lamellar keratoplasty (PALK).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus grades III or IV in the Amsler Krumeich classification.
* Need of surgical procedure
* No endothelial scar
* Best corrected visual acuity <20/40
* Contact lens intolerance
* Imagenological map pachymetric acquisition over 90% at 9 mm corneal diameter

Exclusion Criteria:

* Contraindication for any of the techniques evaluated.
* Requiring additional surgical procedures.
* Diagnostic of other ectasia that were not primary keratoconus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months
  Uncorrected and corrected distance visual acuity

SECONDARY OUTCOMES:
Corneal measurements: pachymetry | 6 months
  Evaluation of the pachymetric maps with a Scheimpflug-Placido device (Sirius). Measurement in microns
Corneal aberrometry: Coma, spherical aberration and trefoil | 6 months
  Evaluation of the corneal aberrations including coma, spherical aberration and trefoil, with a Scheimpflug-Placido device (Sirius)
Corneal measurements: anterior and posterior elevation | 6 months
  Evaluation of the elevation (anterior and posterior), maps with a Scheimpflug-Placido device (Sirius). Measurement in diopters
Corneal measurements: keratometries. | 6 months
  Evaluation of the keratometric map with a Scheimpflug-Placido device (Sirius). Measurement in diopters

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Graue Hernandez, MD, MsC, Study Director — Instituto de Oftalmologia Conde de Valenciana